CLINICAL TRIAL: NCT07186088
Title: Study on the Therapeutic Efficacy of Different Repeated Low-Intensity Red Light Devices and Different Usage Frequencies for Adult Myopia Treatment
Brief Title: Therapeutic Efficacy of Different Repeated Low-Intensity Red Light Devices and Different Usage Frequencies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruihua Wei (Other)
Collaborators: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Ruihua Wei, Professor, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025YK-54
Record Dates: First submitted 2025-08-31; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Laser Group (Experimental): Use Eyerising (RS-200-2A), 1 time,2 times or 3 times a day
  Interventions: Device: Eyerising RS-200-2A
- The LED Group (Experimental): Use Airdoc (Sky-n1201), 2 times a day
  Interventions: Device: Airdoc Sky-n1201

INTERVENTIONS:
Device: Eyerising RS-200-2A — Eyerising RS-200-2A,1 time,2 times, 3 times a day
  Arms: The Laser Group
Device: Airdoc Sky-n1201 — Eyerising RS-200-2A,2 times a day
  Arms: The LED Group

SUMMARY:
To explore the effectiveness and safety of repeated exposure to repeated low-intensity red light

DETAILED DESCRIPTION:
The experiment will be divided into two phases. In the first phase, the subjects will be randomly grouped using laser equipment and LED equipment, and each group will be exposed to the red light twice a day for one month. The second stage involves self-comparison of the laser equipment, with the usage frequencies being once a day and three times a day.

To explore the effectiveness and safety of repeated exposure to repeated low-intensity red light in different devices and frequencies, as well as its impact on the axial length, spherical equivalent refraction and choroidal thickness of myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old, gender not limited; Obtained informed consent.

Exclusion Criteria:

* Obvious strabismus and amblyopia
* With congenital eye disease, such as congenital cataract, congenital retinal disease
* Secondary myopia (such as premature retinopathy or other eye diseases in infants and children caused secondary myopia), or myopia combined with systemic syndrome (such as Marfan syndrome)
* Had internal eye surgery (such as cataract extraction, intraocular lens implantation, anti-glaucoma surgery, etc.)
* Refractive medium opacity (such as corneal disease, crystal opacity, etc.)
* Bnormal intraocular pressure and clinical significance (IOP <10 mmHg or IOP>21mmHg or binocular IOP difference ≥5mmHg)
* Fundus chorioretinopathy (except for high myopia fundus degenerative changes) or other intraocular diseases
* Optic nerve damage or congenital optic nerve dysfunction
* Can not be regularly checked
* The adjustment range is less than 8D or obvious near difficulties
* Other reasons researchers think it is not suitable for inclusion in researchers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Axial length | From enrollment to the end of treatment up to 7 months

SECONDARY OUTCOMES:
Spherical equivalent | From enrollment to the end of treatment up to 7 months
Choroidal thickness | From enrollment to the end of treatment up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Wei, Principal Investigator — Tianjin Medical University Eye Hospital, Tianjin, Tianjin 120120 Recruiting
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No